CLINICAL TRIAL: NCT02804828
Title: Beyond Benefits of Q10: Mitochondrial Cocktail for Gulf War Illness
Brief Title: Mitochondrial Cocktail for Gulf War Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Beatrice Golomb, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: GW140146
Record Dates: First submitted 2015-11-17; First posted 2016-06-17 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Gulf War Syndrome; Persian Gulf Syndrome; Mitochondrial Disorders
MeSH Terms: conditions — Persian Gulf Syndrome; Mitochondrial Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Design study is followed by Crossover to open label treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Dietary Supplement: Individualized mitochondrial cocktail
- Arm 2 (Sham Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Individualized mitochondrial cocktail — Nutrient cocktail comprising: thiamine, nicotinamide, pantothenic acid, riboflavin, L-carnitine, alpha lipoic acid, CoQ10, vitamin C, vitamin E, and omega 3 fatty acids (Cod Liver Oil).
  Arms: Arm 1
Dietary Supplement: Placebo — 6 months for the double-blind phase
  Arms: Arm 2

SUMMARY:
The purpose of this study is to develop preliminary evidence, such as effect size and variance estimates, to guide successful conduct of a properly-powered clinical trial to assess the benefit of a mitochondrial cocktail (incorporating individualization of treatment) in Gulf War illness (GWI).

DETAILED DESCRIPTION:
See below.

ELIGIBILITY:
Inclusion Criteria:

* Meet symptom criteria for Gulf War illness with BOTH the Centers for Disease Control and Prevention (CDC) Criteria (persistent symptoms in at least 2 of 3 designated symptom domains of fatigue/sleep, mood/cognition, and musculoskeletal) and Kansas Criteria (score a moderate or severe rating in at least 3 of the 6 symptom domains of fatigue, pain, neurological/cognitive/mood, skin, GI and respiratory).

Exclusion Criteria:

* Have conditions like multiple sclerosis or lupus that can produce similar symptoms and be confused for Gulf War illness.
* Participating in a concurrent treatment trial.
* Unwilling or unable to comply with the treatment protocol
* Failed run-in; do not take at least 80% of run-in medications

Min Age: 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Mean change in single item General Self-Rated Health Visual Analog Scale from baseline | 0, 3, 6 months (double-blind phase)
Percent improved on Gulf War Illness Modified Lower Extremity Performance Score/timed chair rises | 6 months (double-blind phase)
Number of symptoms (out of 20 on the UCSD Symptom Score Survey) showing more favorable change (trend or effect) on active treatment vs. placebo | 0, 3, 6 months (double-blind phase)
Mean change of CoQ10 and Vitamin E levels, comparing active treatment to placebo | 6 months (double-blind phase)

SECONDARY OUTCOMES:
Assessment of summed symptom score (sum of ratings for UCSD GWI symptom index) | 6, 9, 12 months
  Secondary measures will incorporate assessment of summed symptom score (sum of ratings for UCSD GWI symptom index) at primary endpoint time point. We will assess at additional time points (9, 12 month) and will assess effects stratified by sex; by dominant ethnicity; and by use of medications that can affect levels or disposition of supplement components (e.g. statin use).

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT02804828/ICF_000.pdf